CLINICAL TRIAL: NCT02933606
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study of BNC210 in Adults With Post-Traumatic Stress Disorder (PTSD).
Brief Title: Phase II Study of BNC210 in PTSD
Acronym: RESTORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNC210.007
Record Dates: First submitted 2016-09-01; First posted 2016-10-14 (Estimated); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: Yes

ARMS (4):
- BNC210 600 mg b.i.d. (Experimental): Suspension administered orally for 12 weeks.
  Interventions: Drug: BNC210
- BNC210 300 mg b.i.d. (Experimental): Suspension administered orally for 12 weeks.
  Interventions: Drug: BNC210
- BNC210 150 mg b.i.d. (Experimental): Suspension administered orally for 12 weeks.
  Interventions: Drug: BNC210
- Placebo b.i.d. (Placebo Comparator): Suspension administered orally for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNC210
  Arms: BNC210 150 mg b.i.d.; BNC210 300 mg b.i.d.; BNC210 600 mg b.i.d.
Drug: Placebo
  Arms: Placebo b.i.d.

SUMMARY:
This is a randomized, double-blind, placebo-controlled study, evaluating the effects of BNC210 versus placebo on the symptoms of Post-Traumatic Stress Disorder, as measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).

The secondary objectives of the study are to evaluate the effects of BNC210 on anxiety, depression, global functioning and patient reported outcomes in patients with PTSD. Safety and tolerability of BNC210 will also be assessed. Study participants will receive 12 weeks of blinded treatment followed by a 3 week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated informed consent.
* Male or female between 18 and 70 years of age, inclusive.
* Diagnosed with current PTSD as defined by the CAPS-5 for DSM-5.
* Currently not using any psychiatric medications except for:

  * No more than one selective serotonin reuptake inhibitor (SSRI) (fluvoxamine is excluded) or serotonin noradrenaline reuptake inhibitor (SNRI) within the licensed prescribing dose range. Subjects must have been on a stable dose for at least 3 months prior and through Screening, with the intent to remain on the same dose through to Week 16.
  * As needed (PRN) use of benzodiazepines (BZD) at a frequency not exceeding 2 days per week in the 3 months prior to Screening. The total dose must not exceed 30 mg/day in diazepam equivalents.
* Subjects not currently receiving psychotherapy except long term supportive counseling or subjects that have received intensive regular psychotherapy for a minimum of three months prior to Screening.
* Females of childbearing potential must have a negative serum pregnancy. Females not of childbearing potential must be postmenopausal. Sterilized male patients must be at least 1 year post-vasectomy to be considered of non-child bearing potential. Females and males of childbearing potential must agree to use two effective methods of contraception.

Key Exclusion Criteria

* Current and ongoing exposure to the trauma that caused the PTSD.
* Failed more than three trials of antidepressant medication(s) prescribed for the treatment of PTSD. Each trial must have lasted at least 6 weeks to be considered a failed attempt. A trial that was terminated due to intolerability or side effects does not constitute a failed attempt.
* The use of psychiatric medications within 2 weeks of Screening except for SSRIs, SNRIs or limited PRN BZD use as per inclusion criterion 4. Restricted psychiatric medications include (but are not limited to) antidepressants not allowed by inclusion criterion 4, antianxiety drugs (except limited BZD use per inclusion criterion 4), mood stabilizers, stimulants, antipsychotics, hypnotics and acetylcholinesterase inhibitors.
* History of significant traumatic brain injury.
* Depression as measured by Montgomery-Äsberg depression scale (MADRS) rating > 23.
* Bipolar and psychotic disorders as identified at Screening using the MINI International Neuropsychiatry Interview (V7.0) (M.I.N.I).
* A score ≥ 7 on the McLean Screening Instrument for Borderline Personality Disorder (MSI-BPD) at Screening.
* History of seizure disorders, uncontrolled sleep apnoea or severe neurologic disease.
* Increased risk of suicide, defined as:

  * Any previous suicide attempt disclosed by the participant at Screening using the Columbia Suicide Severity Rating Scale (C-SSRS).
  * Any suicidal ideation with intent (yes to item 4 and / or 5) or suicidal behavior in the past year, as captured at Screening using the C-SSRS.
  * A score > 4 on item 10 of the MADRS at Screening.
* The use of alprazolam or flunitrazepam within 3 months of Screening.
* Any clinically significant abnormalities in laboratory test results, vitals signs, or ECG at Screening.
* Positive result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) at Screening.
* Any moderate to severe substance use disorder (any type) in the 12 months prior to Screening as identified by the DSM-5 using the M.I.N.I (V7.0).
* Current Australian serving Defense personnel or any member of the US military currently serving on active duty.
* Participants involved with ongoing insurance or workplace claims that in the opinion of the Investigator are likely to have an impact on the mental health, presentation or capacity of the patient to engage in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (20):
  - Oceanside, California
  - Rancho Mirage, California
  - Redlands, California
  - Riverside, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lauderhill, Florida
  - North Miami, Florida
  - Oakland Park, Florida
  - Orlando, Florida
  - Hoffman Estates, Illinois
  - Overland Park, Kansas
  - New Bedford, Massachusetts
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Canton, Ohio
  - Memphis, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
- Australia (5):
  - Penrith, New South Wales
  - Auchenflower, Queensland
  - Toowong, Queensland
  - Elizabeth Vale, South Australia
  - St Kilda, Victoria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 193 participants were enrolled into the study and randomized to one of the 4 treatment arms. However, 1 participant withdrew from the study prior to beginning treatment with study IP and hence is not included in the overall number of 192 participants who received study IP and for which post-baseline assessments were performed.
Period: Overall Study
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Started | 49 | 48 | 47 | 49
Completed | 33 | 39 | 33 | 30
Not Completed | 16 | 9 | 14 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d. | Total
Number analyzed (Participants) | 48 | 48 | 47 | 49 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1 | 0 | 2
  Between 18 and 65 years | 46 | 48 | 46 | 49 | 189
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 31 | 30 | 112
  Male | 23 | 22 | 16 | 19 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 16 | 11 | 8 | 10 | 45
  White | 30 | 35 | 36 | 34 | 135
  More than one race | 1 | 1 | 2 | 3 | 7
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 41 | 38 | 161
  Australia | 7 | 7 | 6 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (CAPS-5), Total Symptom Severity Score
Description: Investigator-rated PTSD symptom severity.
  The range for the Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (CAPS-5)Total Symptom Severity Score is 0-80, with a higher score meaning a higher severity of disease.
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 15.26 [11.2 to 19.3] | 16.62 [12.3 to 20.9] | 19.76 [15.5 to 24.0] | 14.57 [9.8 to 19.4]

2. Secondary Outcome: Post-Traumatic Stress Disorder (PTSD) Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (PCL-5).
Description: Self-reported PTSD symptom severity.
  The range for the Post-Traumatic Stress Disorder (PTSD) Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (PCL-5) Symptom Severity Score is 0-80, with a higher score meaning a higher severity of disease.
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 25.02 [19.1 to 31.0] | 20.99 [15.3 to 26.7] | 29.97 [23.5 to 36.4] | 24.65 [17.8 to 31.5]

3. Secondary Outcome: Montgomery- Åsberg Depression Rating Scale (MADRS).
Description: Depression severity.
  The range for the Montgomery- Åsberg Depression Rating Scale (MADRS) is 0-60, with a higher score meaning a higher severity of disease.
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 9.48 [6.7 to 12.3] | 10.25 [7.7 to 12.8] | 12.16 [9.4 to 14.9] | 8.94 [6.1 to 11.8]

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A).
Description: Anxiety severity.
  The range for the Hamilton Anxiety Rating Scale (HAM-A) is 0-56, with a higher score meaning a higher severity of disease.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 9.03 [6.6 to 11.5] | 9.94 [7.6 to 12.3] | 10.55 [8.1 to 13.0] | 7.94 [5.3 to 10.6]

5. Secondary Outcome: Clinical Global Impressions - Severity Scale (CGI-S).
Description: Clinician's assessment of global symptom severity using the Clinical Global Impressions - Severity Scale (CGI-S).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 33 | 39 | 33 | 30
Participants
  Normal, not at all ill | 10 | 5 | 5 | 10
  Borderline mentally ill | 5 | 3 | 6 | 6
  Mildly ill | 8 | 16 | 8 | 5
  Moderately ill | 9 | 13 | 9 | 7
  Markedly ill | 1 | 2 | 3 | 1
  Severely ill | 0 | 0 | 2 | 1
  Among the most extremely ill patients | 0 | 0 | 0 | 0

6. Secondary Outcome: Clinical Global Impressions - Improvement Scale (CGI-I).
Description: Clinician's assessment of global symptom improvement using the Clinical Global Impressions - Improvement Scale (CGI-I).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 33 | 39 | 33 | 30
Participants
  Very Much Improved/Much Improved | 22 | 23 | 15 | 19
  Other | 11 | 16 | 18 | 11

7. Secondary Outcome: Patient Global Impressions - Severity Scale (PGI-S).
Description: Self-reported global symptom severity using the Patient Global Impressions - Severity Scale (CGI-S).
Time Frame: 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 33 | 39 | 33 | 30
Participants
  Normal | 11 | 6 | 6 | 10
  Mild | 8 | 21 | 14 | 13
  Moderate | 12 | 11 | 9 | 3
  Severe | 2 | 1 | 4 | 4

8. Secondary Outcome: Patient Global Impression - Improvement Scale (PGI-I).
Description: Self-reported global symptom improvement using the Patient Global Impression - Improvement Scale (PGI-I).
Time Frame: 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 33 | 39 | 33 | 30
Participants
  Very Much/Much Improved | 17 | 20 | 18 | 20
  Other | 16 | 19 | 15 | 10

9. Secondary Outcome: Assessment of Quality of Life (AQoL-8D).
Description: Quality of Life.
  The range for the Assessment of Quality of Life (AQoL-8D) score is 35-176, with a higher score meaning a lower quality of life.
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 77.95 [71.4 to 84.5] | 76.79 [70.3 to 83.3] | 85.47 [78.0 to 93.0] | 81.05 [73.3 to 88.9]

10. Secondary Outcome: Social Functioning: Sheehan Disability Scale (SDS).
Description: Social functioning.
  The range for the Total Score on the Sheehan Disability Scale (SDS) is 0-30, with a higher score meaning a higher degree of impairment.
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 8.84 [6.2 to 11.5] | 6.66 [4.0 to 9.3] | 10.32 [7.5 to 13.1] | 8.47 [5.3 to 11.7]

11. Secondary Outcome: Sleep Monitoring: Pittsburgh Sleep Quality Index (PSQI).
Description: Sleep quality and duration.
  The range for the Pittsburgh Sleep Quality Index (PSQI) score is 0-21, with a higher score meaning a worse level of sleep quality
Time Frame: 12 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
score on a scale | 8.80 [7.5 to 10.1] | 8.83 [7.6 to 10.1] | 9.15 [7.7 to 10.6] | 8.00 [6.4 to 9.6]

12. Secondary Outcome: CANTAB (Cambridge Neuropsychological Test Automated Battery) Cognitive Assessment
Description: The CANTAB global composite score is based on the Z scores for CANTAB outcome measures (PAL first attempt memory score (PALFAMS), PAL total errors adjusted (PALTEA), SWM between errors (SWMBE), SWM strategy (SWMS), RVP A' prime (RVPA), RVP median latency (RVPMDL). Specifically, the global composite score of cognitive function is as follows: CANTAB global composite score of cognitive function = (ZPALFAMS + ZPALTEA + ZSWMBE + ZSWMS + ZRVPA + ZRVPMDL) /8 (higher is better)
  A Z-score of 0 represents the population mean. A Z-score above 0 indicates cognition higher than the population mean and Z-score below 0 indicates cognition lower than the population mean
Time Frame: 12 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Composite Z score
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
Number analyzed (Participants) | 48 | 48 | 47 | 49
Composite Z score | 0.06 [-0.1 to 0.2] | 0.12 [0.0 to 0.2] | 0.18 [0.1 to 0.3] | 0.02 [-0.1 to 0.2]

ADVERSE EVENTS:
Time Frame: 15 Weeks
Arm/Group | BNC210 600 mg b.i.d. | BNC210 300 mg b.i.d. | BNC210 150 mg b.i.d. | Placebo b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/48 | 0/47 | 1/49
Other Adverse Events (participants affected / at risk) | 31/48 | 42/48 | 30/47 | 45/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNC210 600 mg b.i.d. (N=48) | BNC210 300 mg b.i.d. (N=48) | BNC210 150 mg b.i.d. (N=47) | Placebo b.i.d. (N=49)
Acute Abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Liver Function Tests (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNC210 600 mg b.i.d. (N=48) | BNC210 300 mg b.i.d. (N=48) | BNC210 150 mg b.i.d. (N=47) | Placebo b.i.d. (N=49)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 6 (8) | 4 (4) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (5) | 2 (3) | 6 (9)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 3 (9) | 10 (15) | 4 (4) | 12 (17)
Dizziness (Nervous system disorders) | 2 (2) | 3 (7) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3) | 6 (6) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (5)
Viral Infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (5) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
BNC210 suspension that is dependent on concomitant food intake did not achieve expected exposure levels in the trial participants. However, a planned pharmacometrics analysis established a model of CAPS-5 scores versus plasma exposure and predicted a target exposure for future trials (O'Connor S., SOBP Conference Poster, 2019). A new tablet formulation is being evaluated in a second BNC210 Phase 2 PTSD trial (NCT04951076) and substantially higher exposures are expected in the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02933606/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT02933606/SAP_001.pdf